CLINICAL TRIAL: NCT00168220
Title: Predictors of Drug Hypersensitivity in HIV Infected Subjects
Status: Withdrawn | Type: Observational
Why Stopped: Insufficient recruitment
Sponsor: The Alfred (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Monash University (Other)
Responsible Party: Principal Investigator, Jennifer Hoy, Professor Jennifer Hoy, The Alfred
Other Study IDs: 113/05
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: HIV Infections; Hypersensitivity
Keywords: Treatment Experienced; HIV
MeSH Terms: conditions — HIV Infections; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — plasma, DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Drug hypersensitive group: HIV positive patients with a history of a Hypersensitivity Reaction to the antiretroviral medications Nevirapine, Abacavir or Efavirenz
- Drug tolerant group: HIV positive patients selected based on drug exposure greater than 2 weeks and tolerance to to Abacavir or Nevirapine.

SUMMARY:
A case-control study to look at hypersensitive and tolerant individuals matched for HLA genetic predisposition, when considering predictors of drug hypersensitivity.The study aims to identify the immunological factors increasing the risk of drug reactions in HIV positive individuals.

DETAILED DESCRIPTION:
1. To determine in a case control study clinical parameters associated with drug HSR to abacavir, nevirapine and efavirenz in HIV infected subjects.
2. To measure functional and numerical differences in DC populations and responses to TLR ligands in patients with HSR and tolerant subjects sharing genetic markers for susceptibility to HSR.
3. Identify the role of different DC populations in the development of abacavir reaction by mixing and depletion studies in sensitized subjects and in in vitro assays for abacavir hypersensitivity.
4. To measure T cell parameters including T cell viability in culture, and expression of fas and fasL on blood mononuclear cells in HIV infected controls and HSR patients.
5. To measure blood T cell populations including drug reactive T cells and T regulatory cells in tolerant and reactive subjects with genetic susceptibility to Abacavir and Nevirapine HSR.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected patients on treatment with the drugs Efavirenz, Nevirapine, or Abacavir.
* Age over 18 Cases are those who have had a hypersensitivity reaction, and controls are those who have had no reaction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infection, exposed to antiretroviral treatment, either tolerant or hypersensitive to treatment
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Paul Cameron, Dr, Principal Investigator — The Alfred
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia